CLINICAL TRIAL: NCT01536457
Title: Data Analysis of a Randomized, Double-Blind, Placebo- Controlled Study of Gastroesophageal Reflux Disease Therapy (Lansoprazole; Solutab™) in the Management of Childhood Asthma
Brief Title: Reflux Disease Therapy in the Management of Childhood Asthma-data Entry and Analysis Only
Status: Completed | Type: Observational
Sponsor: Children's Center for Digestive Health Care (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BG-LAN-2011
Record Dates: First submitted 2011-12-29; First posted 2012-02-22 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Asthma; Gastroesophageal Reflux Disease
Keywords: asthma; children; gastroesophageal reflux; retrospective; data analysis
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There have been a number of studies which attribute causality between reflux disease and asthma. In addition, clinicians typically treat chronic asthmatics with high dose acid suppressing medications (e.g. lansoprazole). However, clinical trials only recently have shed some light on this dilemma, with recent studies suggesting that the association is not as clear. This "retrospective" analysis of a prospective study which treated mod-severe asthmatics with lansoprazole or placebo will enter the collected raw data into a database, then perform statistical analyses to determine if children with asthma treated with acid suppression improved their asthma compared to those receiving placebo.

DETAILED DESCRIPTION:
Asthma and gastroesophageal reflux disease (GERD) are common disorders, which are usually non-lethal and both have high morbidity and healthcare costs. Asthma occurs in about 4% - 7% of the US population, and about one-third of active asthmatics are children. There is no universally accepted definition of asthma; it may be regarded as a diffuse, obstructive lung disease with 1) hyper-reactivity of the airways to a variety of stimuli (e.g., acid refluxate via direct exposure and indirect mechanisms; i.e., vagal innervation pathways) and 2) a high degree of reversibility of the obstructive process, which may occur either spontaneously or as a result of treatment. Gastroesophageal reflux (GER) symptoms, which often result in GERD, occur daily in approximately 7% - 20% of the United States adult population; yet population-based studies defining the prevalence of GERD in ambulatory pediatric populations do not exist. Conversely, recent hospital-based data demonstrate that GERD, the intra- and supra-esophageal disease which occurs as a result of GER, is a common pediatric condition resulting in 4% of pediatric hospital discharges across the country. Therefore, asthma and GERD are both common diseases that often appear to co-exist. Moreover, the co-existence of asthma and GERD is far more frequent than chance association. GERD symptoms, although usually mild, occur in up to 65% - 77% of asthmatics. In addition, GERD is common in asthmatics, and is often "silent", i.e. lacking typical symptoms of heartburn. Thus, studies which characterize the relationship between these two conditions and more importantly, interventions which may impact positively on both are critically needed. Moreover, there is data to suggest that both GERD and asthma are life-long conditions that may have childhood origins. A major unanswered question is whether severity or frequency of asthma is related to the response to anti-reflux treatment.

It is also known that acute intermittent reflux, while not meeting established criteria for pathologic GER, can precipitate cough and presumably bronchospasm. Although 1 in 5 asthmatics use bronchodilators to treat symptoms which are interpreted as episodes of heartburn, it is not clear if they are treating bronchospasm or esophageal symptoms. Therefore, one of the aims of this trial was to see if we could demonstrate a significant response to acid-suppression therapy in a group of poorly controlled childhood asthmatics using the number of asthma exacerbations as outcome variables. If there is a causal link between GERD and poor asthma control, one would expect that treatment of GERD would improve asthma. The Cochrane review of evidence-based medicine concluded as follows: "In subjects who had both asthma and GER 51, treatment for GER did not produce a consistent improvement in asthma symptom A subgroup of subjects was reported to gain benefit but it appears difficult to predict responders. At present it is not possible to recommend medical treatment of GER as a means to control asthma. The Cochrane database analysis went on to recommend that "…future research is warranted to examine the effects of therapy for GER on asthma control. Additionally, "…a parallel group, randomized placebo controlled trial (RCT) using a proton pump inhibitor for up to 6 months would be appropriate. Such trials should include assessment and standardized reporting of asthma symptoms, quality of life, lung function, symptom and asthma medication diary, and an assessment of the effects of therapy on GER". Moreover, if GERD and asthma are both lifelong conditions, then one might speculate that overall improvement in health outcomes in adulthood can be achieved by successful detection and intervention in the pediatric age group. Therefore, results from a randomized placebo, controlled treatment trial such as the one we completed and have yet to analyze can surely achieve major health benefit for both children and adults suffering from asthma and GERD, and ultimately change clinical practice that will result in a reduction of the overall public health burden incurred by these chronic human conditions.

It is important for the Institutional Review Board Committee to recognize that the actual "clinical trial" part of the study is complete. This IRB proposal is being submitted to perform perhaps the most critical aspect of the study; the data entry of all of the raw data into secure electronic databases, and then the statistical analysis and interpretation - the final step which we feel the patients and their parents are eager to have completed, and one which we hope will have significant impact in the scientific community - advancing the science behind understanding the relationship between asthma and GERD. More importantly, we feel that by completing the objectives of this new concept proposal - analyzing and interpreting the data obtained in the clinical trial, we will prove our hypothesis - that the treatment of GERD in moderate to severe childhood asthmatics will actually help asthma outcomes - thereby demonstrating that childhood is the critical period in which to intervene in modifying and successfully altering the natural history of these two devastating, chronic diseases with life-long morbidity and healthcare impact (i.e. asthma and GERD).

The actual clinical trial which has been completed is the first investigator initiated trial for the principal investigator and the co-investigators. After IRB approval was obtained IRB #1107-2005, the study enrolled its first patient in March of 2006 and the last patient in December of 2008. The study was also registered with www.clinical trials.gov on October 11, 2005. A Data Safety and Monitoring Board (DSMB) was chartered and formed and met a total of 2 times with one final meeting to be arranged. An external study monitor performed monitoring visits during the first year of the study in order to assure proper protocol compliance, regulatory compliance and study procedure conductance.

The study was completed largely due to the incredible efforts of the GPPA coordinators and Co-investigator. At present, the study is closed, no more patients are being enrolled, and as mentioned, all patients have either completed the study, withdrawn (early termination) or dropped out of the study due to lack of ability to follow up. The study currently retains its "blind" in that all of the raw data has been collected, all of the data remains in source documents (i.e. CRFs) but the data has not been entered into the secure electronic database, and subsequently, thus, no data analysis has occurred, interpretation provided or study conclusions drawn.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were enrolled in the study, "Randomized, Double-blind, Placebo Controlled Study of Gastroesophageal Reflux Disease Therapy (Lansoprazole; Solutab™) in the Management of Childhood Asthma" will be entered into this database. Only these patients will be included in this study, all other patients will be excluded.

Exclusion Criteria:

* Patients who were not enrolled in the study, "Randomized, Double-blind, Placebo Controlled Study of Gastroesophageal Reflux Disease Therapy (Lansoprazole; Solutab™) in the Management of Childhood Asthma" will not be included in this study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a retrospective study. The study will simply be taking data collected during a prospective study and analyzing that data. There will be no subjects enrolled in this retrospective study. The subjects enrolled in the prospective study were children, ages 4 to 11 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations in the treatment group | Over 21 months
  This is a retrospective study. We will be entering data collected in a prospective clinical trial and then analyzing such data to determine if intervention with acid suppression, lansoprazole improves the number of asthma exacerbation in a one year period compared to those receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Gold, M.D., Principal Investigator — Children's Center for Digestive Health Care
Locations (1):
- Children's Center for Digestive Health Care, Atlanta, Georgia, United States